CLINICAL TRIAL: NCT06944574
Title: Sleep Intervention Swiss Elite Athletes
Acronym: SISEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Sport Magglingen (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-02076; PT00P1_199093 / 1 (Other: Swiss National Science Foundation)
Record Dates: First submitted 2025-04-02; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-10

CONDITIONS: Sleep Problems
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (one arm only, repeated measure design) (Experimental)
  Interventions: Behavioral: Guided online intervention

INTERVENTIONS:
Behavioral: Guided online intervention — The intervention combines a one-hour in-person workshop with a four-week app-based program tailored to elite athletes. The workshop focuses on sleep education and individual motivation setting. Athletes then complete seven self-paced audio modules via the "7-Schläfer" app, covering strategies to improve sleep quality. Weekly reminder emails reinforce motivation. Unlike other interventions, this program is fully integrated into the elite sport context, emphasizes behavioral change through personalized goal-setting, and includes no therapist contact, ensuring scalability. No control group is included in this one-arm pre-post design.

SUMMARY:
Background and Rationale Elite athletes frequently experience sleep disturbances due to factors like irregular schedules, travel, and pre-competition stress. Despite the critical role of sleep in physical recovery and mental health, many athletes fail to meet sleep quality recommendations. While sleep interventions have shown promise in improving sleep outcomes, their effects on mental health-especially in athlete populations-remain underexplored. This study investigates the impact of a 4-week app-based sleep intervention, preceded by a workshop, on both sleep and mental health outcomes in Swiss elite athletes.

Objective To evaluate whether a brief, structured sleep intervention improves sleep quality and mental health in elite athletes and to identify perceived facilitators and barriers to intervention success.

Design A single-center, one-arm pre-post intervention study with four time points (baseline, pre-intervention, post-intervention, and 2-month follow-up). No control group is used due to practical constraints.

Participants 16 elite athletes (sport soldiers) enrolled in the Swiss recruit school. All participants are adults and proficient in German.

Intervention

A one-hour sleep workshop covering the importance of sleep and motivation-setting.

A four-week app-based program ("7-Schläfer") with seven audio modules (approx. 30 minutes each), completed flexibly by participants.

Outcomes

Primary outcomes include:

Sleep quality and disturbances

Mental health (depression, anxiety, well-being)

Data will be collected via REDCap using validated questionnaires. After the intervention, individual interviews will gather qualitative feedback.

Analysis Quantitative data will be analyzed using repeated measures ANOVA. Focus group data will be analyzed thematically.

Significance The study aims to provide practical, scalable insights into how sleep-focused interventions can improve athlete well-being and inform recommendations for sport organizations.

DETAILED DESCRIPTION:
1. Background and Rationale Elite athletes often suffer from sleep disturbances due to high training loads, frequent travel, jet lag, pre-competition stress, and irregular routines. Poor sleep negatively affects cognitive function, immune response, recovery, and overall performance. It is also strongly associated with mental health challenges including anxiety, depression, and psychological distress.

   Although interventions such as sleep hygiene education and sleep extension strategies show promise in improving subjective sleep quality, there is limited evidence on their long-term effectiveness or impact on mental health in elite athlete populations. Moreover, few studies examine what elements of sleep interventions athletes perceive as most helpful or what barriers they face.

   This study seeks to close these gaps by evaluating the short- and long-term effects of a structured sleep intervention on sleep quality and mental health in elite Swiss athletes, with additional qualitative data on user experience.
2. Study Objectives Primary Objective To determine whether a 4-week sleep intervention improves sleep quality and mental health (depression, anxiety, and well-being) in elite athletes.

   Hypotheses

   The intervention will reduce sleep disturbances and improve sleep quality.

   The intervention will enhance mental health outcomes, including reduced symptoms of depression and anxiety and improved well-being.

   Secondary Objectives To explore participant experiences, including perceived facilitators, barriers, and the most helpful components of the intervention.
3. Study Design

   This is a national, single-center, one-arm pre-post intervention study using a within-subjects design. It includes four measurement time points:

   T0: Baseline

   T1: Pre-intervention

   T2: Post-intervention

   T3: Two-month follow-up
4. Participants Sample Size: 16 elite athletes from the recruit school (sport soldiers).

   Inclusion Criteria:

   Enrolled in the recruit school

   Elite athlete status

   Sufficient understanding of German

   Exclusion Criteria:

   Insufficient German to engage with the app

   All participants are adults capable of providing informed consent.
5. Intervention Component 1: Workshop A one-hour in-person workshop focused on the importance of sleep for physical and mental performance, sleep hygiene strategies, and goal setting. Participants identify personal motivations, which are later used to encourage adherence.

   Component 2: App-Based Sleep Program ("7-Schläfer") Participants complete 7 modules (approx. 30 minutes each) over four weeks. Modules include guided audio exercises and psychoeducation about sleep. Participants can take private notes, which are not accessed by the research team. Weekly reminder emails with personalized motivational cues are sent to enhance engagement.

   Participation in the intervention is free of charge. The app is provided at no cost and without data sharing.
6. Outcomes and Measurements

   Validated questionnaires will be used:

   Sleep Quality: Visual analog scale (1 item)

   Sleep Disturbance: Insomnia Severity Index (ISI, 7 items)

   Well-Being: MHC-SF (14 items)

   Depression: PHQ-9 (9 items)

   Anxiety: GAD-7 (7 items)

   Participants also report demographic data, sport type, training intensity, and adherence (module completion and perceived usefulness). Post-intervention, optional focus groups (2 groups of 6-9 athletes) explore facilitators, barriers, and perceived effectiveness.
7. Data Collection and Management All data is collected through REDCap. Only three project staff members have access. Identifying data is stored separately and pseudonymized.
8. Statistical Analysis Repeated measures ANOVA will assess within-subject changes across the four time points. Power analysis determined that 24 participants are needed for moderate effect detection. To account for attrition, 30 athletes will be recruited.

   Qualitative data from focus groups will be analyzed using thematic analysis. Gender will be included as a control variable.

   Missing data will be handled using multiple imputation. Participants must complete at least baseline and post-intervention assessments to be included in analysis.
9. Ethics and Risk Assessment The study is categorized as minimal risk (ClinO, Art. 61, Cat. A). No vulnerable populations are included. Ethical risks are low and primarily involve potential distress when reflecting on sleep habits. Participants are provided with mental health resources and may contact the research team or sport psychology services at any time.
10. Monitoring and Safety A trained monitor from the Swiss Federal Institute of Sport will conduct site visits at initiation, mid-study, and study close-out. Serious Adverse Events will be reported per ClinO requirements. No radiation, invasive procedures, or vulnerable groups are involved.
11. Registration and Dissemination The study will be registered with SNCTP and ClinicalTrials.gov. Results will be published open access and anonymized data will be made publicly available after project completion.
12. Funding Funded by the Swiss National Science Foundation (project number PT00P1_199093 / 1). There are no financial or personal conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

elite athlete participating in the recruit school (sport soldiers), understanding German because the content of the App is only available in German

Exclusion Criteria:

not understanding German good enough to understand the content of the App

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Sleep problems | The ISI was administered at four time points: (1) baseline, (2) pre-intervention (4 weeks later, immediately before intervention), (3) post-intervention (6 weeks after pre-intervention), and (4) follow-up (2 months after post-intervention).
  The Insomnia Severity Index (ISI, Gerber et al., 2016) was used to assess the severity of sleep problems. The ISI consists of seven items, evaluating difficulties with falling asleep, staying asleep, subjective sleep quality, the impact of sleep disturbances on daily life, and worries about sleep problems in the previous two weeks. Participants rated each item on a 5-point scale ranging from 0 (not at all) to 4 (very much). A total sleep problem score was calculated by summing all item responses. Higher values indicate more sleep problems.

SECONDARY OUTCOMES:
Depression | The PHQ-9 was administered at four time points: (1) baseline, (2) pre-intervention (4 weeks later, immediately before intervention), (3) post-intervention (6 weeks after pre-intervention), and (4) follow-up (2 months after post-intervention).
  The 9-item Patient Health Questionnaire (PHQ-9, Kroenke et al., 2001) was used to assess depressive symptoms in the two preceding weeks. The PHQ-9 asks participants to self-assess nine problems (e.g., "I had little interest or pleasure in doing things") on a 4-point scale ranging from not at all (0) to nearly every day (3). A total depression score was obtained by summing all item responses. Higher scores indicate more depressive symptoms.
Anxiety | The GAD-7 was administered at four time points: (1) baseline, (2) pre-intervention (4 weeks later, immediately before intervention), (3) post-intervention (6 weeks after pre-intervention), and (4) follow-up (2 months after post-intervention).
  The 7-item General Anxiety Disorder (GAD-7, Spitzer et al., 2006; Spitzer et al., 1999) was used to assess anxiety symptoms in the two preceding weeks. The GAD-7 asks participants to self-assess seven core symptoms of generalized anxiety disorder (e.g., "I had not been able to stop or control worrying") on a 4-point scale ranging from not at all (0) to nearly every day (3). A total anxiety score was obtained by summing all item responses. Higher scores indicate more anxiety symptoms.
Well-being | The MHC-SF was administered at four time points: (1) baseline, (2) pre-intervention (4 weeks later, immediately before intervention), (3) post-intervention (6 weeks after pre-intervention), and (4) follow-up (2 months after post-intervention).
  To assess well-being, we used the 14-item Mental Health Continuum Short Form (MHC-SF, Lamers et al., 2011). The MHC-SF comprises three subscales: emotional well-being (three items; e.g., "During the past month, how often did you feel satisfied with life?"); social well-being (five items; e.g., "During the past month, how often did you feel that you had something important to contribute to society?"); and psychological well-being (six items; e.g., "During the past month, how often did you feel that you had experiences that challenged you to grow and become a better person?"). Items are rated on a 6-point scale ranging from never (1) to every day (6), and mean scores are calculated for the three subscales and the total scale. Higher score indicate greater well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Federal Institute of Sport Magglingen, Magglingen, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Small study sample with elite athletes, sharing data cannot garantee anonymity of participants